CLINICAL TRIAL: NCT01220115
Title: A 3-year, Prospective, Non-interventional, Multicenter Registry in Sickle Cell Disease Patients
Brief Title: A 3-year, Prospective, Non-interventional, Multicenter Registry in Sickle Cell Disease (SCD) Patients
Acronym: FISCO
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CICL670AUS38
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2015-05

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; iron over load
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No treatment: Patients aged 2 to less than 12
- No treatment patients aged 12 to less than 18: Patients aged 12 to less than 18
- No treatment Patients greater than 18 years: patients greater than 18 years

SUMMARY:
A long term observational study in sickle cell disease will enhance the understanding of the disease patterns, current transfusion practices, treatments and outcomes in sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with HbSS, HbS/beta-thalassemia and HbSC
* Age > 2 years old.
* Written informed consent by the patient or legal guardians, and pediatric assent where indicated.

Exclusion Criteria:

* Patients with Sickle Cell trait (HbAS) are not eligible for the study
* Patient or legal guardians unable or unwilling to give consent, or pediatric assent where indicated.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Sickle cell disease age 2 years and older
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Document current treatment patterns, natural history and outcomes in patients with sickle cell disease | up to 5 years

SECONDARY OUTCOMES:
Data collection | up to 5 years
  Collection of the following data:Current therapies used for the treatment of SCD Current transfusion practices, Difference in treatments between pediatric and adult patients, Use of chelation therapies, Frequency and types of crises including Frequency of hospitalizations, Incidence of end organ damage (caridac, renal, pulmonary,liver), Quality of life assessed by PedsQL TM Pediatric Quality of Life Inventory for patients 2- <18 years old and SF-36® Health Survey for patients 18 years old and older
Measure Sickle cell crisis and hospitalizations | up to 5 years
  To evaluate whether patients on regular transfusion protocol have fewer crisis and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- United States (42):
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Children's Hospital Oakland (CHO), Oakland, California
  - Children's Hospital of Orange County Sickle Cell Disease Center, Orange, California
  - Rady Children's Hopsital / UC San Diego University Hospital Sickle Cell Disease Center, San Diego, California
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Howard University, Washington D.C., District of Columbia
  - Broward Oncology Associates, P.A., Fort Lauderdale, Florida
  - Miami Children's Hospital, Miami, Florida
  - Innovative Medical Research, Miami, Florida
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Central Tampa Hematology and Oncology Associates, Tampa, Florida
  - St. Joseph Children's Hospital, Tampa, Florida
  - University of Illinois at Chicago, Dept of Pediatrics, Chicago, Illinois
  - Abington Hematology Oncology Associates, Inc, Oak Lawn, Illinois
  - Tulane University School of Medicine, New Orleans, Louisiana
  - LSU Department of Pediatrics Children's Hospital, New Orleans, Louisiana
  - Johns Hopkins University Division of Hematology, Baltimore, Maryland
  - Oncology-Hematology Associates, P.A., Clinton, Maryland
  - Children's Hospital Boston - Harvard, Boston, Massachusetts
  - Boston Comprehensive Sickle Cell Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Missouri Child Health, Division of Pediatric Hematology/Oncology, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - New York Methodist Hospital Dept of Med/Sickle Cell Program, Brooklyn, New York
  - Interfaith Medical Center-Comprehensive Sickle Cell Program, Brooklyn, New York
  - Cohen Children's Medical Center of NY (CCMC), New Hyde Park, New York
  - Center for Children's Cancer & Blood Disorders, Syracuse, New York
  - Presbyterian Hospital Pediatric Sickle Cell Program, Charlotte, North Carolina
  - Ohio Region VI Sickle Cell Program, Akron, Ohio
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Medical University of SC-Pediatric Sickle Cell Center, Charleston, South Carolina
  - M. Francisco Gonzalez, M.D., P.A., Columbia, South Carolina
  - Diggs-Kraus Sickle Cell Center, Memphis, Tennessee
  - Meharry Comprehensive Sickle Cell Center, Nashville, Tennessee
  - Sickle Cell Disease and Hemoglobinopathy Clinic Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Baylor College of Medicine-Texas Children's Hospital, Houston, Texas
  - Peninsula Cancer Institute, Newport News, Virginia